CLINICAL TRIAL: NCT02501434
Title: A Blind-adjudication Multi-center Phase II Randomized Clinical Trial of Continuous Low-dose Intravenous Heparin Therapy in Coiled Low-grade Aneurysmal Subarachnoid Hemorrhage Patients With Significant Hemorrhage Burden
Brief Title: Aneurysmal Subarachnoid Hemorrhage Trial RandOmizing Heparin
Acronym: ASTROH
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Robert F. James (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Robert F. James, Professor of Neurosurgery, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10550
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Neurobehavioral Manifestations; Vasospasm, Intracranial; Intracranial Aneurysm; Heparin-induced Thrombocytopenia Type II
Keywords: aneurysmal subarachnoid hemorrhage; unfractionated heparin; neurobehavioral manifestations; delayed ischemic neurological deficits; cerebral aneurysm; coil embolization; Montreal Cognitive Assessment
MeSH Terms: conditions — Subarachnoid Hemorrhage; Neurobehavioral Manifestations; Vasospasm, Intracranial; Intracranial Aneurysm | interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Control (No Intervention): Standard of Care
- LDIVH (Unfractionated Heparin) (Experimental): Continuous Low-Dose IV Unfractionated Heparin Infusion
  Interventions: Drug: Continuous Low-Dose IV Unfractionated Heparin Infusion

INTERVENTIONS:
Drug: Continuous Low-Dose IV Unfractionated Heparin Infusion — Continuous intravenous infusion of a low-dose unfractionated heparin drip
  Other Names: Heparin; Unfractionated Heparin; Heparin drip; IV Heparin
  Arms: LDIVH (Unfractionated Heparin)

SUMMARY:
A Blind-adjudication Multi-center Phase II Randomized Clinical Trial of Continuous Low-dose Intravenous Heparin Therapy in Coiled Low-grade Aneurysmal Subarachnoid Hemorrhage Patients with Significant Hemorrhage Burden. - STUDY IS TEMPORARILY SUSPENDED WITH PLAN TO RESUME SOON. NO SAFETY CONCERNS

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety and clinical effect of a continuous low-dose intravenous unfractionated heparin (LDIVH) infusion for the prevention of aneurysmal subarachnoid hemorrhage (aSAH) induced neurocognitive dysfunction and other delayed neurological deficits.

Additionally, increased blood and CSF levels of certain inflammatory biomarkers (IL-6, hsCRP, etc) have been correlated to aSAH patients with poor clinical outcomes. Unfractionated heparin (UFH) has known anti-inflammatory actions. As a result, a secondary objective of this study will be to evaluate whether LDIVH can reduce blood and CSF inflammatory biomarkers levels compared to controls and whether there is any association between inflammatory biomarker levels and cognitive outcomes in aSAH.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 70 years
2. Historical modified Rankin Scale Score 0-1
3. Aneurysmal subarachnoid hemorrhage caused by a ruptured saccular aneurysm confirmed by catheter angiography that is repaired by endovascular coil embolization. Initiation of the coil embolization procedure should occur within 48 hours from the time of the aneurysm rupture (ictus). In patients where the exact time of the ictus is uncertain, a reasonable estimate of the time of ictus may be assigned. This reasonable time estimate should be considered likely accurate to within hours of the true unknown time.
4. Quality of aneurysm embolization is interpreted to be Raymond-Roy Score of 1 (Complete) or 2 (Residual Neck) indicating that the aneurysm is adequately secured. A tiny amount of contrast in the body of the aneurysm is acceptable as long as the physician considers the aneurysm secured and to NOT represent a Raymond-Roy Score of 3 (Residual Aneurysm).
5. WFNS grade 1 or 2 as assessed after repair of the aneurysm during screening but prior to randomization. A patient who presents with a WFNS greater than 2 who then improves with resuscitation, ventriculostomy, or time is acceptable.
6. The pre-repair, admission head CT demonstrates an aSAH bleed pattern of "thick and diffuse" or "thick and focal" hemorrhage within the subarachnoid basal cisterns measuring ≥ 4 mm in the short axis and ≥ 20 mm in the long axis which is consistent with a modified Fisher grade 3 or 4. Intraventricular hemorrhage is acceptable. Enrollable patients must NOT have a parenchymal hemorrhage greater than 10 cc. Please refer to diagram below for examples. The hemorrhage location should be substantially within the supratentorial space and not isolated to the infratentorial space.
7. The location of the aneurysm should be the anterior circulation, posterior communicating, OR a basilar terminus (apex). Angiographic location of the aneurysm should be confirmed by catheter digital subtraction angiography (DSA) usually obtained during the coil embolization procedure. Patients with PICA or other posterior circulation aneurysms as the cause of the SAH should not be included because they typically cause primarily infratentorial bleed patterns.
8. Ability to screen the patient and obtain a head CT 2-12 hours after the completion of the coiling procedure and the ability to initiate the study drug 12 ± 8 hours after the completion of aneurysm coiling procedure.
9. After recovering from anesthesia following the aneurysm coiling procedure, the patient must remain a WFNS SAH grade ≤ 2 without evidence of a significant new focal neurological deficit including monoparesis / monoplegia, hemiparesis / hemiplegia, or receptive, expressive or global aphasia. New minor cranial nerve defect without any other new findings is permissible. If an NIHSS score was obtained prior to the aneurysm coiling procedure, a post-coiling (pre-enrollment) NIHSS score must not have increased by ≥ 4 points and GCS score must not be decreased by ≥ 2 points. The clinician at the local site should use their best clinical judgment as to whether a significant neurological decline has occurred due to the procedure.
10. Patient is willing and able to return for study follow-up visits.
11. Patient or their Legally Authorized Representative (LAR) has provided written informed consent.

Exclusion Criteria:

1. Angio-negative SAH.
2. History or imaging suggesting that the current hemorrhage presentation is a recent re-rupture of the aneurysm. Prior sentinel headache with negative CT or prior sentinel headache where the patient did not seek medical attention does not exclude the patient.
3. Surgical Clipping (or plan for clipping) of the ruptured aneurysm or any non- ruptured aneurysm on the same admission.
4. Aneurysm is identified to be traumatic, mycotic, blister or fusiform type by catheter DSA.
5. Any intracranial stent placement or non-coil intra-aneurysmal device where dual- antiplatelet therapy is needed during admission.
6. Patient has additional aneurysm(s) that are untreated and could reasonably be considered a possible alternate cause of the aSAH based on the observed bleeding pattern. Adequate treatment of these aneurysms by coiling embolization would result in the aneurysms no longer causing an exclusion. MRI may be used in some situations to determine that the associated aneurysms did not rupture based on lack of blood seen adjacent to the additional aneurysms.
7. Patient received heparin in any form within the last 100 days prior to current presentation / admission.
8. Thrombocytopenia (platelet count less than 100,000 - assuming clumping has been ruled out as a cause).
9. New intraparenchymal hemorrhage or new infarction larger the 15cc in volume, or significant increased mass effect as seen on the post-coiling, pre-enrollment head CT when compared to baseline admission head CT. New hyperdensity on CT scan related to contrast staining is not an exclusion.
10. Patient has a documented history of heparin induced thrombocytopenia (HIT).
11. Patient developed SAH-induced cardiac stunning prior to enrollment, with an ejection fraction <30%, or requiring IV medications for blood pressure maintenance.
12. Concurrent significant intracranial pathology identified prior to enrollment, including but not limited to, Moyamoya disease, high suspicion or documented CNS vasculitis, severe fibromuscular dysplasia, arteriovenous malformation, arteriovenous fistula, or malignant brain tumor.
13. Thrombolytic therapy within 24 hours prior to enrollment (rtPA, urokinase, etc.)
14. Plan for antiplatelet or oral anticoagulation therapy from the time of the coil embolization procedure until 14 full days after enrollment. Antiplatelet therapy may be resumed after the 14-day window. A single 325 mg Aspirin (or lower dose) given during the coil embolization peri-procedural period is acceptable if this is the local standard of care but should be documented.
15. Concomitant serious or uncontrolled disease such as severe infection, active (non- remission) cancer, severe organ dysfunction (severe heart failure, severe chronic kidney impairment requiring dialysis or severe chronic liver disease) or any coagulopathy (including DIC or bleeding diathesis).
16. Uncontrollable hypertension (>180 systolic and/or >110 diastolic) that is not correctable prior to enrollment.
17. Prior neurological disease/deficit or psychiatric disease that may continue to alter the results of neuropsychological evaluation, such as dementia, Multiple sclerosis, seizure disorder, severe traumatic brain injury, previous ruptured cerebral aneurysm or active major depression. Childhood seizures that have resolved and no longer require treatment are not part of this exclusion criteria.
18. Active Immunosuppression therapy including chronic corticosteroid usage.
19. History of gastrointestinal hemorrhage or major systemic hemorrhage within 30 days (including large flank or large retroperitoneal hematoma due to current admission coiling procedure requiring treatment), hemoglobin less than 6 g/dL, INR ≥1.5 after reversal of anticoagulants.
20. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days.
21. Currently pregnant.
22. Enrollment in another research study that prescribes a therapeutic treatment that differs from the local standard of care, or that would conflict with this study in some other significant fashion. Registries or coil comparison studies are appropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 90-day follow-up visit
  Primary Clinical Outcome Measure- mean score compared between groups
Rate of "Major Bleeding" or "Clinically Relevant Non-Major Bleeding" | Patients will be followed for the duration of the hospital stay; an expected average of 3 weeks
  As defined by the International Society of Thrombosis and Heamostasis (ISTH) Primary Safety Outcome Measure-

SECONDARY OUTCOMES:
Rate of "Major Bleeding" | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
  As defined by the International Society of Thrombosis and Haemostasis (ISTH)
Rate of Type II Heparin Induced Thrombocytopenia (HIT) | Enrollment through 90-day follow-up visit
Rate of Deep Venous Thrombosis (DVT) or Pulmonary Embolism (PE) | Enrollment through 90-day follow-up visit
All Cause - Mortality Rate | Enrollment through 90-day follow-up visit
Incidence of Any Fever (> 38.3 degrees C; > or = 101.0 degrees F) | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
Incidence of multiple fevers (> 2 episodes) | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
Mean daily fever burden | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
  Daily fever burden = Sum of hourly fever burden over 24 hours; Hourly fever burden = Any hourly temperature recording > 37 degrees C - (minus) 37 degrees C; if temperature is less than or equal to 37 degrees C then the hourly fever burden would be zero.
Glasgow Coma Score | Enrollment, post-enrollment days #6, 10, discharge, and 90-day follow-up visit
National Institutes of Health Stroke Scale (NIHSS) | Enrollment, post-enrollment days #6, 10, upon discharge from hospital stay an expected average of about 3 weeks after admission, 90-day follow-up visit
Montreal Cognitive Assessment (MoCA) | Enrollment, post-enrollment days #6, 10, 1 year follow-up
  Mean between groups and rate of MoCA score of 20 or less between groups
Center for Epidemiologic Studies Depression Scale (CES-D) | 90-day follow-up visit and 1-year follow-up visit
Trail Making Test Parts A&B | 90-day follow-up visit
Cerebral Vasospasm | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
  Incidence of moderate and severe radiographic cerebral vasospasm (catheter angiogram, CTA, MRA) or incidence OR moderate and severe vasospasm by transcranial doppler (TCD) criteria
Incidence of clinical cerebral vasospasm requiring rescue therapy | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
  Rescue therapy = vasopressors or endovascular therapy for the purposes of reversing clinical vasospasm; it does not include Triple H (Hyperdynamic Therapy)
Incidence of CT or MRI imaging demonstrating cerebral vasospasm related cerebral infarction | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks
Ordinal Regression Analysis of the modified Rankin Scale score (mRS) | 90-day follow-up visit and 1 year follow-up visit
Relative frequency of "good outcome" as defined by dichotomized mRS score 0-2 | 90-day follow-up visit and 1 year follow-up visit
Barthel Index | 90-day follow-up visit and 1 year follow-up visit
Return to work status | 90-day follow-up and 1 year follow-up visit
Lawton instrumental activities of daily living (IADL) | 90-day follow-up visit and 1 year follow-up visit
Quality of Life in Brain Injury - Overall Scale (QOLIBRI-OS) | 90-day follow-up visit and 1 year follow-up visit
Checklist Individual Strength- Subscale Fatigue (CIS-F) | 90-day follow-up visit and 1 year follow-up visit
Plasma biomarker level (hsCRP) | Enrollment, post-enrollment days #2,4,6,10
Cerebrospinal Fluid (CSF) biomarker level (hsCRP) | Enrollment, post-enrollment days #2,4,6,10
Rate of Serious Adverse Events (SAEs) | From enrollment through 90-Day follow-up visit
  Secondary Safety Outcome Measure

OTHER OUTCOMES:
Subgroup analysis for the following subgroups: (Clinical Site, Gender, Admission CT Hijdra Sum Score <23, WFNS grade, aneurysm location, anterior circulation aneurysm vs posterior circulation aneurysm location, infection requiring antibiotic treatment, | Participants will be followed for the duration of the hospital stay, an expected average of 3 weeks, 90-day follow-visit and 1 year follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Robert F James, MD, Principal Investigator — Indiana University; J Marc Simard, MD, PhD, Principal Investigator — University of Maryland; J Mocco, MD, MSc, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kevin N Sheth, MD, Principal Investigator — Yale University
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Rush University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai Ichan School of Medicine, New York, New York
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data other than through publication or requests to Robert James by other investigators.

REFERENCES:
- [Background] Simard JM, Schreibman D, Aldrich EF, Stallmeyer B, Le B, James RF, Beaty N. Unfractionated heparin: multitargeted therapy for delayed neurological deficits induced by subarachnoid hemorrhage. Neurocrit Care. 2010 Dec;13(3):439-49. doi: 10.1007/s12028-010-9435-1. PMID 20809188
- [Background] Al-Khindi T, Macdonald RL, Schweizer TA. Cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. Stroke. 2010 Aug;41(8):e519-36. doi: 10.1161/STROKEAHA.110.581975. Epub 2010 Jul 1. PMID 20595669
- [Background] Schweizer TA, Al-Khindi T, Macdonald RL. Mini-Mental State Examination versus Montreal Cognitive Assessment: rapid assessment tools for cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. J Neurol Sci. 2012 May 15;316(1-2):137-40. doi: 10.1016/j.jns.2012.01.003. Epub 2012 Jan 26. PMID 22280947
- [Background] Wong GK, Lam SW, Ngai K, Wong A, Mok V, Poon WS. Quality of Life after Brain Injury (QOLIBRI) Overall Scale for patients after aneurysmal subarachnoid hemorrhage. J Clin Neurosci. 2014 Jun;21(6):954-6. doi: 10.1016/j.jocn.2013.09.010. Epub 2013 Nov 9. PMID 24373816
- [Background] Hong CM, Tosun C, Kurland DB, Gerzanich V, Schreibman D, Simard JM. Biomarkers as outcome predictors in subarachnoid hemorrhage--a systematic review. Biomarkers. 2014 Mar;19(2):95-108. doi: 10.3109/1354750X.2014.881418. Epub 2014 Feb 5. PMID 24499240
- [Background] Romero FR, Bertolini Ede F, Figueiredo EG, Teixeira MJ. Serum C-reactive protein levels predict neurological outcome after aneurysmal subarachnoid hemorrhage. Arq Neuropsiquiatr. 2012 Mar;70(3):202-5. doi: 10.1590/s0004-282x2012000300009. PMID 22392113
- [Background] Fountas KN, Tasiou A, Kapsalaki EZ, Paterakis KN, Grigorian AA, Lee GP, Robinson JS Jr. Serum and cerebrospinal fluid C-reactive protein levels as predictors of vasospasm in aneurysmal subarachnoid hemorrhage. Clinical article. Neurosurg Focus. 2009 May;26(5):E22. doi: 10.3171/2009.2.FOCUS08311. PMID 19409001
- [Background] Tosun C, Kurland DB, Mehta R, Castellani RJ, deJong JL, Kwon MS, Woo SK, Gerzanich V, Simard JM. Inhibition of the Sur1-Trpm4 channel reduces neuroinflammation and cognitive impairment in subarachnoid hemorrhage. Stroke. 2013 Dec;44(12):3522-8. doi: 10.1161/STROKEAHA.113.002904. Epub 2013 Oct 10. PMID 24114458
- [Background] Simard JM, Aldrich EF, Schreibman D, James RF, Polifka A, Beaty N. Low-dose intravenous heparin infusion in patients with aneurysmal subarachnoid hemorrhage: a preliminary assessment. J Neurosurg. 2013 Dec;119(6):1611-9. doi: 10.3171/2013.8.JNS1337. Epub 2013 Sep 13. PMID 24032706
- [Background] James RF, Shao EY, Page PS, Nazar RG, Martin LB, Dvorak J, Kanaan HK, Daniels MJ, Craycroft J, Rai SN, Everhart DE, Simard JM. Low-dose IV heparin preserves cognitive function in aneurysmal subarachnoid hemorrhage patients. [Unpublished Data]. Presented at AANS 82nd Annual Scientific Meeting. April 5-9, 2014. San Francisco, CA; Abstract #16572.